# Study protocol: "Biological evolution of HELLP syndrome".

#### I. Introduction:

HELLP syndrome is considered a clinical form of preeclampsia (or toxemia gravidarum), which itself is a severe complication of the second and third trimesters of pregnancy. However, in 15% of cases, it can occur in isolation in the absence of signs of preeclampsia.

It is associated with hemolysis, thrombocytopenia and hepatic cytolysis. The diagnosis and management of HELLP syndrome are still the subject of controversy, and its management depends on two therapeutic attitudes: conservative treatment with close monitoring, or rapid termination of pregnancy, taking into account gestational age and clinical and biological severity.

The aim of this study is to investigate the biological evolution of HELLP syndrome before and after extraction.

### II. Study characteristics

- Type of study: prospective observational
- Study setting: maternal intensive care unit at the Hôpital Mère -Enfant CHU Mohammed VI,
  Marrakech
- Principal investigators: Pr Ahmed Rhassane El Adib/ Pr Essafti Meryem / Dr Nizar Amllah
- Inclusion criteria: Patients admitted to maternal intensive care for complete or incomplete biological HELLP syndrome.
- Exclusion criteria: Patients whose biological profile is explained by another pathology (other microangiopathies, leukemia, etc.).
- Study procedure: The study will not entail any change in patient care, and will proceed as follows:

o Inclusion of patients after informing them of the characteristics of the study and obtaining their consent.

- o Questioning about the various pathological histories.
- o Search for complications according to their clinical picture.
- o Daily collection of biological data.
- o Recording of transfusion events, and administration of corticosteroid therapy according to term.
- o Recording of extraction and analgesia techniques.

## III. Potential dangers to subjects

This study does not involve any risks, since it is based solely on data collection.

# IV. Confidentiality Protection:

Medical data concerning patients is governed by medical secrecy and all data recorded in the information sheet is only identifiable through a numerical identifier assigned to patients at the time of inclusion. As the protection of all medical data is a priority, such data will be identified by a code number (IP) without the use of personal names or initials. These data may be transmitted to the various entities participating in the study under strict conditions of confidentiality.